CLINICAL TRIAL: NCT03544515
Title: Treatment of Peri-implantitis: Clinical Comparison Between Conventional Treatment Versus Conventional Plus Biolase Laser Treatment as a Co-adjuvant
Brief Title: Peri-implantitis Treatment: Clinical Results of Conventional Treatment vs. the Addition of Biolase
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: Biolase Inc (Industry)
Responsible Party: Principal Investigator, Philip Y. Kang, Associate Professor of Dental Medicine, Columbia University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AAAR8727
Record Dates: First submitted 2018-04-30; First posted 2018-06-01 (Actual); Results first posted 2024-08-09 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-07

CONDITIONS: Peri-Implantitis
Keywords: peri-implantitis; laser treatment; Biolase; Er,Cr:YSGG
MeSH Terms: conditions — Peri-Implantitis | interventions — Tooth Exfoliation

STUDY DESIGN:
Intervention Model Description: Double blind randomized clinical trial
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Scaling and use of inactive Er,Cr:YSGG (Sham Comparator): Scaling and debridement with hand scalers and ultrasonic unit together with the application of the Er,Cr:YSGG laser in an inactive fashion
  Interventions: Procedure: Scaling; Device: Inactive Er,Cr:YSGG
- Scaling and use of active Er,Cr:YSGG (Experimental): Scaling and debridement with hand scalers and ultrasonic unit together with the application of the Er,Cr:YSGG laser in an active fashion
  Interventions: Device: Er,Cr:YSGG laser; Procedure: Scaling

INTERVENTIONS:
Device: Er,Cr:YSGG laser — Application of Er,Cr:YSGG in peri-implantitis cases as a coadjutant has shown reduction in the pocket depths and bleeding on probing
  Other Names: Biolase (Biolase, Inc)
  Arms: Scaling and use of active Er,Cr:YSGG
Procedure: Scaling — Scaling and debridement of the implant surface with hand scalers and curettes and an ultrasonic scaling unit (Cavitron -Dentsply Sirona)
Device: Inactive Er,Cr:YSGG — Er,Cr:YSGG laser (inactive form - sham procedure) applied to the surface of the implant
  Arms: Scaling and use of inactive Er,Cr:YSGG

SUMMARY:
The purpose of the study is to observe the effects of two commonly utilized treatment modalities to treat peri-implantitis and to compare the results. The first method of treatment is debridement with curettes and ultrasonic scalers and it represents the traditional approach in the treatment of peri-implantitis. The second method of treatment involves the use of the Biolase laser in addition to the traditional approach of debriding with curettes and ultrasonic scalers. No studies exist comparing these two approaches, and this will serve as a pilot study to explore possible differences. The research hypothesis is that the addition of Er;Cr;YSGG laser is likely to be more effective in removing the microbiota from a rough implant surface, and that this will manifest with improved clinical parameters in subjects that receive this method of treatment.

DETAILED DESCRIPTION:
Peri-implantitis has been defined as an implant restoration with inflamed bleeding gingiva, probing depths around the implant of 5-8mm, bone loss and exposure of threads around the implant (limited to one-third of the threads exposed). The purpose of this study is to determine the benefits of treating peri-implantitis with a closed laser approach known as the "Repair Protocol" using an Er,Cr:YSGG laser compared with traditional non-surgical therapy. Each subject, when determined to fall under the parameters of the study for peri-implantitis, will be randomly assigned to one of two groups: the test Er,Cr:YSGG laser group or the control group.

The study will constitute a human double-blind randomized clinical trial in which both examiners and patients will be blinded to the treatment. In order to ensure the blinding of the patients, the laser will be applied to all implants, although the it will not be activated in the control group. The therapist will be the same person throughout the study while the examiners will be calibrated.

The two groups that will constitute the study and the procedures that will be applied are:

Experimental: Scaling and root planning with an ultrasonic or piezoelectric instrument and hand instrumentation with hand instruments. No prosthetic components will be removed . Application of laser therapy following the specifics of the company.

Control: Scaling and root planning with an ultrasonic or piezoelectric instrument and hand instrumentation with hand instruments. A sham, inactivated laser, treatment will be delivered.

After the treatment, the patients will be followed-up after 1 week, 3, 6 and 9 months. Periapical X-rays will be taken at baseline and 9 months follow-up appointments.

Data to be collected include: Primary outcome measures will include: presence of bleeding on probing, probing depth, and the progression of bone loss around the implant, as measured with bone sounding under local anesthesia and radiographically with the aid of a stent. Secondary outcome measures will include: Gingival index (GI), Plaque Index, mobility, and suppuration.

ELIGIBILITY:
Inclusion Criteria:

* Presence of at least one implant presenting with early to moderate peri-implantitis
* Peri-implantitis defined as an implant restoration with inflamed bleeding gingiva, probing depths around the implant of 5-8mm, bone loss and exposure of threads around the implant (limited to one-third of the threads exposed).
* Medically healthy non-smokers with no previous periodontal treatment other than routine maintenance
* Patients with diabetes were only included if they reported an HbA1C of 7% or less within the past 3 months

Exclusion Criteria:

* Mobility of the implant
* Peri-implantitis treatment rendered in the last 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2019-01-14 (Actual); Primary Completion 2021-08-02 (Actual); Study Completion 2021-08-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Philip Kang, DDS, Principal Investigator — Columbia University College of Dental Medicine
Locations (1):
- Columbia University College of Dental Medicine, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Scaling and Use of Inactive Er,Cr:YSGG | Scaling and Use of Active Er,Cr:YSGG
Started | 16 | 15
Completed | 10 | 13
Not Completed | 6 | 2
Not completed — Didn't complete study follow-up due to pandemic pause in research activity | 4 | 2
Not completed — Lost to Follow-up | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Scaling and Use of Inactive Er,Cr:YSGG | Scaling and Use of Active Er,Cr:YSGG | Total
Number analyzed (Participants) | 16 | 15 | 31
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.19 (9.26) | 62.53 (7.12) | 64.93 (8.49)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 2 | 6
  Male | 12 | 13 | 25
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 16 | 15 | 31
Implant Prosthesis [Number; unit: implants]
  screw-retained | 19 | 8 | 27
  cement-retained | 41 | 20 | 61

OUTCOME MEASURES:

1. Primary Outcome: Change in Probing Depth (PD)
Description: Measured in mm with a manual periodontal probe (UNC-15). Recorded at 6 sites per implant (mesio-buccal and lingual, mid-buccal and lingual, disto-buccal and lingual). The average of all sites for all implants (26 implants in the Inactive Arm; 38 implants in the Active Arm) is reported.
Time Frame: Baseline, 9 months
Population: Analyzed 10 out of 16 subjects who completed the study in the control (inactive) group, and 13 out of 15 subjects who completed the study in the laser (active) group.
Measure: Mean (95% Confidence Interval); unit: mm
Units Other Than Participants: implants
Arm/Group | Scaling and Use of Inactive Er,Cr:YSGG | Scaling and Use of Active Er,Cr:YSGG
Number analyzed (Participants) | 10 | 13
Number analyzed (implants) | 26 | 38
mm | -0.73 [-1.17 to 0.28] | -1.36 [-1.96 to 0.77]

2. Secondary Outcome: Change in Radiographic Bone Loss Around the Implant
Description: Measured with calibrated (taken with a positioning device) peri-apical X-rays. Radiographic bone loss is measured as distance from the platform of the implant to the crest of the bone in the mesial and distal sites. The average of all sites for all implants (26 implants in the Inactive Arm; 38 implants in the Active Arm) is reported.
Time Frame: Baseline, 9 months
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: mm
Units Other Than Participants: impants
Arm/Group | Scaling and Use of Inactive Er,Cr:YSGG | Scaling and Use of Active Er,Cr:YSGG
Number analyzed (Participants) | 10 | 13
Number analyzed (impants) | 26 | 38
mm | 0.02 [-0.56 to 0.61] | 0.05 [-0.80 to 0.91]

3. Secondary Outcome: Mean Change in Percent of Implants That Presented Bleeding on Probing (BoP)
Description: Recorded at 6 sites per implant (mesio-buccal and lingual, mid-buccal and lingual, disto-buccal and lingual). The average of all sites for all implants (26 implants in the Inactive Arm; 38 implants in the Active Arm) is reported.
Time Frame: Baseline, 9 months
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: percentage of bleeding
Units Other Than Participants: implants
Arm/Group | Scaling and Use of Inactive Er,Cr:YSGG | Scaling and Use of Active Er,Cr:YSGG
Number analyzed (Participants) | 10 | 13
Number analyzed (implants) | 26 | 38
percentage of bleeding | -20 [-37 to -2] | -36 [-61 to -1]

4. Secondary Outcome: Presence of Suppuration on Probing
Description: Recorded at 6 sites per implant (mesio-buccal and lingual, mid-buccal and lingual, disto-buccal and lingual). Dichotomic
Time Frame: 9 months
Population: Data was not collected.
Arm/Group | Scaling and Use of Inactive Er,Cr:YSGG | Scaling and Use of Active Er,Cr:YSGG
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Plaque Index (PI): Mean Change in Percent of Implants That Contained Plaque
Description: as for outcome 3
Time Frame: Baseline, 9 months
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: percentage of plaque
Units Other Than Participants: implants
Arm/Group | Scaling and Use of Inactive Er,Cr:YSGG | Scaling and Use of Active Er,Cr:YSGG
Number analyzed (Participants) | 10 | 13
Number analyzed (implants) | 38 | 26
percentage of plaque | -30 [-50 to -8] | -29 [-54 to -2]

6. Secondary Outcome: Mobility: Mean Change in the Clinical Attachment Level (CAL)
Description: CAL is an indicator of the stability of the implant. CAL is measured in mm as distance from the cemento-enamel junction to the gingival margin.
Time Frame: Baseline, 9 months
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: mm
Units Other Than Participants: implants
Arm/Group | Scaling and Use of Inactive Er,Cr:YSGG | Scaling and Use of Active Er,Cr:YSGG
Number analyzed (Participants) | 10 | 13
Number analyzed (implants) | 26 | 38
mm | -1.2 [-1.97 to -0.36] | -0.90 [-1.34 to -0.47]

ADVERSE EVENTS:
Time Frame: Up to 9 months
Arm/Group | Scaling and Use of Inactive Er,Cr:YSGG | Scaling and Use of Active Er,Cr:YSGG
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/13
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/13
Other Adverse Events (participants affected / at risk) | 0/10 | 0/13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-02-23): https://cdn.clinicaltrials.gov/large-docs/15/NCT03544515/Prot_SAP_000.pdf